CLINICAL TRIAL: NCT02258867
Title: A Randomized-Withdrawal, Double-Masked, Placebo-Controlled Study of the Efficacy and Safety of Gevokizumab in Treating Subjects With Behcet's Disease Uveitis
Brief Title: Efficacy and Safety Study of Gevokizumab to Treat Behcet's Disease Uveitis
Acronym: EYEGUARD™-US
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: XOMA (US) LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: X052133
Record Dates: First submitted 2014-10-02; First posted 2014-10-08 (Estimated); Last update posted 2015-12-29 (Estimated); Status verified 2015-12

CONDITIONS: Behcet's Disease Uveitis
Keywords: Uveitis; Behcet's Disease Uveitis; Behcet's Disease
MeSH Terms: conditions — Uveitis; Behcet Syndrome | interventions — gevokizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- Gevokizumab (Experimental)
  Interventions: Drug: Gevokizumab

INTERVENTIONS:
Drug: Placebo — Solution for subcutaneous injection
  Arms: Placebo
Drug: Gevokizumab — Solution for subcutaneous injection
  Arms: Gevokizumab

SUMMARY:
The objective of this study is to assess the efficacy and safety of gevokizumab in treating Behcet's disease uveitis (BDU).

ELIGIBILITY:
Inclusion Criteria:

* Have characteristics of Behcet's disease consistent with International Criteria for Behcet's disease
* Have a documented history of active uveitis with or without retinal vasculitis within the past 12 months
* Best corrected visual acuity (BCVA) >= 20 ETDRS letters in both eyes at baseline
* Effective contraceptive measures

Exclusion Criteria:

* Infectious uveitis and masquerade syndromes
* End stage ocular disease
* History of allergic or anaphylactic reactions to monoclonal antibodies
* Active tuberculosis disease
* History of recurrent infection or predisposition to infection; active ocular infection
* Pregnant or nursing women

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2014-11; Primary Completion 2015-10 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Time to first ocular exacerbation | Randomization through Day 280
  Time to first ocular exacerbation is defined as the number of days from randomization to the first ocular exacerbation.

CONTACTS AND LOCATIONS:
Locations (8):
- United States (8):
  - Santa Ana, California
  - Chicago, Illinois
  - Ellsworth, Maine
  - Cambridge, Massachusetts
  - Royal Oak, Michigan
  - Winston-Salem, North Carolina
  - Fargo, North Dakota
  - Houston, Texas